CLINICAL TRIAL: NCT05683158
Title: Compensatory Kinematic Movement for Reaching Task in Various Directions in After Stroke
Brief Title: Compensatory Kinematic Movements in Various Directions After Stroke
Status: Completed | Type: Observational
Sponsor: University of Valencia (Other)
Collaborators: Ulsan National Institute of Science and Technology (Unknown)
Responsible Party: Principal Investigator, José Casaña Granell, Principal Investigator, University of Valencia
Other Study IDs: Kinematic movements of stroke
Record Dates: First submitted 2022-12-21; First posted 2023-01-12 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Cerebral Stroke; Hemiplegia, Spastic
Keywords: Chronic stroke; Reaching task; Motion capture
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- chronic stroke: The subject consisted of the physician's confirmation of chronic hemiplegia onset ≥ 6 months Mini-mental state examination≥25 Biceps ≤2, Triceps≤2 Ability to Sit on a chair alone FMA upper extremity score ≥ 21points, FMA upper extremity score ≤ 66 points The symptom is mild or moderate level (MAS≤2) and can sit alone. The subject reaches to target by affected arm in 3 directions(medial_45, forward_90 and lateral_135 degrees)
- Healthy: Matching aged people, not having neurological system or orthopedic disease on Upper extremity.
  The subject reaches to target by non-dominant arm in 3 directions(medial_45, forward_90 and lateral_135 degrees)

SUMMARY:
This is cross-sectional study. By comparing kinematic analysis between stroke and healthy subjects in various directions, this investigation analyzes the compensatory kinematic movement for reaching task in stroke survivors

DETAILED DESCRIPTION:
After Institutional Review Board approval, It recruits 2 groups. one group is elderly and another group is stroke survivors. the stroke group that meets the criteria. Another group is age matching of the stroke and not having an orthopedic or neurological disease. Participants of all the groups are assessed for kinematic by motion capture During reaching arm(affected side; stroke group, non-dominant side; healthy group) in 3 directions(medial_45, forward_90 and lateral_135 degrees). Retroreflective markers are placed on 11 anatomical place (3th metacarpal joint, both acromion, elbow lateral and medial epicondyle, lateral and medial styloid process, xyphoid process, sternum, C7, T4). Participants reach to a bell as quickly as possible in three directions. The subject reach to a bell 5 times in each direction and assess clinical evaluation such as Fugl Meyer Assessment, Postural Assessment Scale, Modified Ashworth Scale, shoulder-elbow range of motion and Trunk Instability scale.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria used in the randomized controlled trials were as follows:

Stroke

* Subject consisted of the physician's confirmation of chronic hemiplegia
* onset ≥ 6 months
* Mini-mental state examination≥25
* Biceps ≤2, Triceps≤2
* Ability to Sit on a chair alone
* FMA upper extremity score ≥ 21 points, FMA upper extremity ≤ 66 points

Healthy

* Age of matching the stroke group
* Absence of neurological disease and orthopedic disease

Exclusion Criteria:

Stroke

* Biceps>2, Triceps>2
* Flaccid
* Neglect syndrome
* Have neurological disease and orthopedic disease
* Lack of coordination

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruit research participants from the healthy group of 61 participants at the gym for the disabled of Ulsan city and Ulsan national institute of science and technology. Another group of 35 patients who enter the largest gym for the disabled of Ulsan city.
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jóse Casaña Granell, PhD, Principal Investigator — University of Valencia; Joaquin Calatayud Villalba, PhD, Principal Investigator — University of Valencia; Sang Hoon Kang, PhD, Principal Investigator — Ulsan National Institute of Science and Technology
Locations (1):
- Ulsan National Institute of Science and Technology, Ulsan, Ulju, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alt Murphy M, Murphy S, Persson HC, Bergstrom UB, Sunnerhagen KS. Kinematic Analysis Using 3D Motion Capture of Drinking Task in People With and Without Upper-extremity Impairments. J Vis Exp. 2018 Mar 28;(133):57228. doi: 10.3791/57228. PMID 29658937
- [Background] Wu CY, Liing RJ, Chen HC, Chen CL, Lin KC. Arm and trunk movement kinematics during seated reaching within and beyond arm's length in people with stroke: a validity study. Phys Ther. 2014 Jun;94(6):845-56. doi: 10.2522/ptj.20130101. Epub 2014 Jan 30. PMID 24481598
- [Background] Machado LR, Heathcock J, Carvalho RP, Pereira ND, Tudella E. Kinematic characteristics of arm and trunk when drinking from a glass in children with and without cerebral palsy. Clin Biomech (Bristol). 2019 Mar;63:201-206. doi: 10.1016/j.clinbiomech.2019.03.011. Epub 2019 Mar 19. PMID 30925379
- [Background] Lobo-Prat J, Font-Llagunes JM, Gomez-Perez C, Medina-Casanovas J, Angulo-Barroso RM. New biomechanical model for clinical evaluation of the upper extremity motion in subjects with neurological disorders: an application case. Comput Methods Biomech Biomed Engin. 2014 Aug;17(10):1144-56. doi: 10.1080/10255842.2012.738199. Epub 2012 Nov 27. PMID 23181596
- [Background] Hsieh YW, Liing RJ, Lin KC, Wu CY, Liou TH, Lin JC, Hung JW. Sequencing bilateral robot-assisted arm therapy and constraint-induced therapy improves reach to press and trunk kinematics in patients with stroke. J Neuroeng Rehabil. 2016 Mar 22;13:31. doi: 10.1186/s12984-016-0138-5. PMID 27000446
- [Background] Cirstea MC, Levin MF. Compensatory strategies for reaching in stroke. Brain. 2000 May;123 ( Pt 5):940-53. doi: 10.1093/brain/123.5.940. PMID 10775539
- [Background] Levin MF, Michaelsen SM, Cirstea CM, Roby-Brami A. Use of the trunk for reaching targets placed within and beyond the reach in adult hemiparesis. Exp Brain Res. 2002 Mar;143(2):171-80. doi: 10.1007/s00221-001-0976-6. Epub 2002 Jan 8. PMID 11880893
- [Background] Adamovich SV, Archambault PS, Ghafouri M, Levin MF, Poizner H, Feldman AG. Hand trajectory invariance in reaching movements involving the trunk. Exp Brain Res. 2001 Jun;138(3):288-303. doi: 10.1007/s002210100694. PMID 11460767
- [Background] Dean CM, Shepherd RB. Task-related training improves performance of seated reaching tasks after stroke. A randomized controlled trial. Stroke. 1997 Apr;28(4):722-8. doi: 10.1161/01.str.28.4.722. PMID 9099186
- [Background] Dean C, Shepherd R, Adams R. Sitting balance I: trunk-arm coordination and the contribution of the lower limbs during self-paced reaching in sitting. Gait Posture. 1999 Oct;10(2):135-46. doi: 10.1016/s0966-6362(99)00026-0. PMID 10502647
- [Background] Thrane G, Sunnerhagen KS, Murphy MA. Upper limb kinematics during the first year after stroke: the stroke arm longitudinal study at the University of Gothenburg (SALGOT). J Neuroeng Rehabil. 2020 Jun 15;17(1):76. doi: 10.1186/s12984-020-00705-2. PMID 32539738
- [Background] Cirstea MC, Mitnitski AB, Feldman AG, Levin MF. Interjoint coordination dynamics during reaching in stroke. Exp Brain Res. 2003 Aug;151(3):289-300. doi: 10.1007/s00221-003-1438-0. Epub 2003 Jun 19. PMID 12819841
- [Background] Schwarz A, Veerbeek JM, Held JPO, Buurke JH, Luft AR. Measures of Interjoint Coordination Post-stroke Across Different Upper Limb Movement Tasks. Front Bioeng Biotechnol. 2021 Jan 28;8:620805. doi: 10.3389/fbioe.2020.620805. eCollection 2020. PMID 33585418

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician's confirmation of chronic hemiplegia with ≥ 6 months onset and the healthy group consisted of individuals without any history of neurological or orthopedic diseases. The participants was enrolled from August, 2022 to June, 2023 at the gym for the disabled of Ulsan city and Ulsan national institute of science and technology
Pre-assignment Details: All of the subjects of 96 enrolled participants were inclusion criteria
Period: Overall Study
Arm/Group | Chronic Stroke | Healthy
Started | 35 | 61
Completed | 35 | 61
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: To determine the sample size, the G*Power software was utilized, incorporating an effect size (d) of 1.9, alpha level of 0.05, and power of 0.8. A sample size of six individuals per group was considered sufficient to achieve adequate statistical power, which are α ≤ 0.05, power = 0.8, and β = 0.2. Consequently, a suitable number of participants were recruited, considering a comparison of 35 individuals in the stroke group and 61 individuals in the healthy group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Chronic Stroke | Healthy | Total
Number analyzed (Participants) | 35 | 61 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 18 | 30
  >=65 years | 23 | 43 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.80 (13.81) | 68.61 (7.23) | 68.67 (10.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 32 | 49
  Male | 18 | 29 | 47
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  South Korea | 35 | 61 | 96
Fugl-Meyer Assessment (FMA) [Median (Inter-Quartile Range); unit: units on a scale] — Inclusion criteria: FMA upper extremity score ≥ 21 points (In sitting position, the sum of each subtotal score is 66 (maximum) and the minimum is 0. Subscales were summed to compute a total score Cutoff scores defined 21 ~ 50: moderate, 51~66: mild
  1) Reflex activity_max 4 score, 2) Volitional movement within synergies_ max 18, 3) Volitional movement mixing synergies_ max 6, 4) Volitional movement with little or no synergy_ max 6, 5) Normal reflex activity_max 2, 6) Wrist movement_ max 10, 7) Hand movement with grasp_ max 14, 8) coordination/speed_max 6.
  units on a scale | 51 [32 to 64] | 66 [66 to 66] | 66 [61.25 to 66]

OUTCOME MEASURES:

1. Primary Outcome: Differences in Spatial Measurements of Trunk Dislocation Components During 3-directional Bell-reaching Task Between Healthy Subjects and Stroke Patients
Description: Trunk dislocation (reaching phase in millimetre; mm) in reaching task. The measurements are detected in 3 directions (Forward_90, Lateral_135, Medial_45 degree). Participants reach to a bell as quickly as possible. 3rd joint is calculated for quantitative measurements.
Time Frame: 1 time (Baseline)
Population: The population analyzed enrolled all participants with inclusion criteria between chronic stroke and healthy
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Chronic Stroke | Healthy
Number analyzed (Participants) | 35 | 61
millimeter
  Trunk dislocation (mm)_Forward | 272.44 (88.63) | 221.24 (71.37)
  Trunk dislocation (mm)_Lateral | 288.14 (90.99) | 253.50 (74.54)
  Trunk dislocation (mm)_Medial | 274.83 (88.31) | 230.76 (80.51)
Statistical Analysis 1: Comparison: Chronic Stroke vs Healthy; To determine the sample size, the G*Power software was utilized, incorporating an effect size (d) of 1.9, alpha level of 0.05, and power of 0.8. A sample size of six individuals per group was considered sufficient to achieve adequate statistical power, which are α ≤ 0.05, power = 0.8, and β = 0.2; Test type: Other; p < .001, ANOVA; Mean Difference (Net) = 1.71, Standard Error of Mean 0.28 — Mean difference between two groups of movement unit in forward direction
Statistical Analysis 2: Comparison: Chronic Stroke vs Healthy; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < .001, ANOVA; Mean Difference (Net) = 0.44, Standard Error of Mean 0.12 — Statistics difference among forward, ipsilateral and contralateral directions in within group

2. Primary Outcome: Differences in Spatial Measurements of Elbow and Shoulder Angle Components During 3-directional Bell-reaching Task Between Healthy Subjects and Stroke Patients
Description: Elbow extension and shoulder flexion angle (degree) in reaching task. The measurements are detected in 3 directions (Forward_90, Lateral_135, Medial_45 degree). Participants reach to a bell as quickly as possible. 3rd joint is calculated for quantitative measurements.
Time Frame: 1 time (Baseline)
Population: The population analyzed enrolled all participants with inclusion criteria between chronic stroke and healthy
Measure: Mean (Standard Deviation); unit: Degree
Arm/Group | Chronic Stroke | Healthy
Number analyzed (Participants) | 35 | 61
Degree
  Elbow extension_Forward | 132.27 (20.53) | 131.97 (9.26)
  Elbow extension_Lateral | 133.70 (19.44) | 135.20 (13.20)
  Elbow extension_Medial | 127.04 (24.93) | 127.46 (12.31)
  Shoulder flexion_Forward | 131.49 (19.39) | 123.29 (18.12)
  Shoulder flexion_Lateral | 130.95 (21.43) | 128.64 (13.39)
  Shoulder flexion_Medial | 135.00 (18.55) | 123.67 (13.80)

3. Primary Outcome: Differences in Temporal Measurements of Movement Unit Components During 3-directional Bell-reaching Task Between Healthy Subjects and Stroke Patients
Description: Movement units are quantified by counting velocity peaks during the reaching task. A movement unit is defined as a velocity profile segment between a local minimum and the following maximum velocity that exceeds 20 mm/s, with a minimum time interval of 150 ms between subsequent peaks. This measure represents the smoothness of movement, where fewer movement units indicate smoother motion The measurements are detected in 3 directions (Forward_90, Lateral_135, Medial_45 degree). Participants reach to a bell as quickly as possible. 3rd joint is calculated for quantitative measurements.
Time Frame: 1 time (Baseline)
Population: The population analyzed enrolled all participants with inclusion criteria between chronic stroke and healthy
Measure: Mean (Standard Deviation); unit: number of peaks
Arm/Group | Chronic Stroke | Healthy
Number analyzed (Participants) | 35 | 61
number of peaks
  Movement unit_Forward | 4.47 (2.17) | 3.18 (0.80)
  Movement unit_Lateral | 5.02 (2.60) | 2.63 (0.67)
  Movement unit_Medial | 4.11 (1.94) | 2.66 (0.76)

4. Primary Outcome: Differences in Temporal Measurements of Hand Movement Time Components During 3-directional Bell-reaching Task Between Healthy Subjects and Stroke Patients
Description: The period from hand tangential velocity movement onset to offset was the total time (entire time of reach and return phase [second]). The period when the tangential velocity exceeded 10% of its peak was termed hand movement onset, whereas that when the tangential velocity stayed below 10% of its peak was termed hand movement offset.
  The measurements are detected in 3 directions (Forward_90, Lateral_135, Medial_45 degree). Participants reach to a bell as quickly as possible. 3rd joint is calculated for quantitative measurements.
Time Frame: 1 time (Baseline)
Population: The population analyzed enrolled all participants with inclusion criteria between chronic stroke and healthy
Measure: Mean (Standard Deviation); unit: second
Arm/Group | Chronic Stroke | Healthy
Number analyzed (Participants) | 35 | 61
second
  Total time_Forward | 3.42 (1.13) | 2.09 (0.44)
  Total time_Lateral | 3.49 (1.21) | 2.07 (0.40)
  Total time_Medial | 3.26 (1.02) | 1.98 (0.37)

5. Primary Outcome: Differences in Temporal Measurements of Hand Velocity Components During 3-directional Bell-reaching Task Between Healthy Subjects and Stroke Patients
Description: Tangential velocity was computed for the hand marker's velocity. Peak elbow angular velocity (rad/s) during elbow extension were measured The measurements are detected in 3 directions (Forward_90, Lateral_135, Medial_45 degree). Participants reach to a bell as quickly as possible. 3rd joint is calculated for quantitative measurements.
Time Frame: 1 time (Baseline)
Population: The population analyzed enrolled all participants with inclusion criteria between chronic stroke and healthy
Measure: Mean (Standard Deviation); unit: rad/s
Arm/Group | Chronic Stroke | Healthy
Number analyzed (Participants) | 35 | 61
rad/s
  Elbow angular velocity_Forward | 45.66 (31.21) | 75.40 (39.87)
  Elbow angular velocity_Lateral | 44.04 (29.60) | 76.47 (43.44)
  Elbow angular velocity_Medial | 53.74 (37.60) | 79.15 (38.79)

6. Primary Outcome: Differences in Temporal Measurements of Elbow Extension Acceleration Components During 3-directional Bell-reaching Task Between Healthy Subjects and Stroke Patients
Description: Acceleration (rad/s2) during elbow extension was measured The measurements are detected in 3 directions (Forward_90, Lateral_135, Medial_45 degree). Participants reach to a bell as quickly as possible. 3rd joint is calculated for quantitative measurements.
Time Frame: 1 time (Baseline)
Population: The population analyzed enrolled all participants with inclusion criteria between chronic stroke and healthy
Measure: Mean (Standard Deviation); unit: rad/s2
Arm/Group | Chronic Stroke | Healthy
Number analyzed (Participants) | 35 | 61
rad/s2
  Elbow angular acceleration_Forward | 344.75 (261.56) | 628.85 (270.49)
  Elbow angular acceleration_Lateral | 321.28 (199.17) | 542.96 (281.04)
  Elbow angular acceleration_Medial | 396.78 (320.56) | 722.87 (280.19)

7. Primary Outcome: Difference of the Components Temporal Measurements Between Healthy and Stroke
Description: Tangential velocity was computed for the hand marker's velocity. The period when the tangential velocity exceeded 10% of its peak was termed hand movement onset, whereas that when the tangential velocity stayed below 10% of its peak was termed hand movement offset. Peak hand velocity (mm/s) was analyzed.
  The measurements are detected in 3 directions (Forward_90, Lateral_135, Medial_45 degree). Participants reach to a bell as quickly as possible. 3rd joint is calculated for quantitative measurements.
Time Frame: 1 time (Baseline)
Population: The population analyzed enrolled all participants with inclusion criteria between chronic stroke and healthy
Measure: Mean (Standard Deviation); unit: mm/s
Arm/Group | Chronic Stroke | Healthy
Number analyzed (Participants) | 35 | 61
mm/s
  Hand velocity_Forward | 944.52 (610.70) | 805.28 (324.31)
  Hand velocity_Lateral | 1003.22 (634.69) | 822.19 (270.58)
  Hand velocity_Medial | 1015.06 (675.14) | 1188.89 (497.50)

8. Secondary Outcome: Comparison of Fugl-Meyer Assessment Scores Between Chronic Stroke Patients and Healthy
Description: Related Fugl-Meyer Assessment score(dependent) to predictors(independent) in three directions.
  In sitting position, the sum of each subtotal score is 66 (maximum) and the minimum is 0. Subscales were summed to compute a total score. Cutoff scores defined 0~20: severe, 21 ~ 50: moderate, 51~66: mild
  1) Reflex activity_max 4 score, 2) Volitional movement within synergies_ max 18, 3) Volitional movement mixing synergies_ max 6, 4) Volitional movement with little or no synergy_ max 6, 5) Normal reflex activity_max 2, 6) Wrist movement_ max 10, 7) Hand movement with grasp_ max 14, 8) coordination/speed_max 6.
Time Frame: Baseline
Population: The population analyzed enrolled all participants with inclusion criteria between chronic stroke and healthy
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Chronic Stroke | Healthy
Number analyzed (Participants) | 35 | 61
score on a scale | 51 [32 to 64] | 66 [66 to 66]

9. Other Pre Specified Outcome: Comparison of Modified Ashworth Scale Between Chronic Stroke Patients and Healthy Controls
Description: Scoring for Biceps
  * MAS 0: No increase in tone
  * MAS 1: slight increase in tone giving a catch when slight increase in muscle t-tone, manifested by the limb was moved in flexion or extension.
  * MAS 1+: slight increase in muscle tone, manifested by a catch followed by minimal resistance throughout (ROM )
  * MAS 2: more marked increase in tone but more marked increased in muscle tone through most limb easily flexed
  * MAS 3: considerable increase in tone, passive movement difficult
  * MAS 4: limb rigid in flexion or extension The Modified Ashworth Scale (MAS) ranges from 0 to 4, where higher scores indicate more severe spasticity/increased muscle tone. A score of 0 represents normal muscle tone, while 4 represents the most severe level of spasticity.
Time Frame: Baseline
Population: The population analyzed enrolled all participants with inclusion criteria between chronic stroke and healthy
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Chronic Stroke | Healthy
Number analyzed (Participants) | 35 | 61
score on a scale | 2 [0 to 2] | 0 [0 to 0]

10. Other Pre Specified Outcome: Range of motion_Health Status Chronic Stroke
Description: Shoulder and elbow joint range of motion
  * Shoulder flexion, adduction, abduction, external rotation, internal rotation
  * Elbow flexion, extension
Time Frame: Baseline
Population: The population analyzed enrolled all participants with inclusion criteria between chronic stroke and healthy
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Chronic Stroke | Healthy
Number analyzed (Participants) | 35 | 61
degree
  Shoulder flexion | 161.46 (22.16) | 179.02 (7.68)
  Shoulder abduction | 149.57 (34.11) | 179.26 (5.76)
  Shoulder adduction | 44.77 (8.82) | 50.00 (0)
  Shoulder external rotation | 71.86 (19.18) | 89.51 (2.36)
  Shoulder internal rotation | 76.94 (19.79) | 87.70 (8.09)
  Elbow flexion | 139.63 (7.29) | 144.18 (3.05)
  Elbow extension | 1.94 (5.26) | 0 (0)

11. Other Pre Specified Outcome: Trunk Impairment Scale(TIS)_Health Status Chronic Stroke
Description: The Trunk Impairment Scale (TIS) for stroke has a total score of 23 points, with higher scores indicating better trunk control ability. TIS components:
  Static sitting balance - 7 points Dynamic sitting balance - 10 points Coordination - 6 points 23 points = Optimal trunk control ability (normal performance of all items) 0 points = Minimal trunk control ability (unable to perform) Static sitting balance Dynamic sitting balance Co-ordination
Time Frame: 1 time(Baseline)
Population: The population analyzed enrolled all participants with inclusion criteria between chronic stroke and healthy
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Chronic Stroke | Healthy
Number analyzed (Participants) | 35 | 61
score on a scale | 14 [11 to 20] | 23 [23 to 23]

12. Other Pre Specified Outcome: Postural Assessment Scale for Stroke(PASS)_Health Status Chronic Stroke
Description: The Postural Assessment Scale for Stroke (PASS) evaluates postural control in stroke patients, with scores ranging from 0-36 points, where higher scores indicate better functional recovery.
  1) Sitting without support 2,3) Standing with(without) support 4,5) Standing on (non)paretic leg 6) Supine to affected side lateral 7) Supine to non-affected side lateral 8) Supine to sitting up on the edge of the table 9) Sitting on the edge of the table to supine 10) Sitting to standing up 11) Standing up to sitting down 12) Standing, picking up a pencil from the floor
Time Frame: Baseline
Population: The population analyzed enrolled all participants with inclusion criteria between chronic stroke and healthy
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Chronic Stroke | Healthy
Number analyzed (Participants) | 35 | 61
score on a scale | 33 [32 to 34] | 36 [36 to 36]

13. Other Pre Specified Outcome: Fugl_Meyer Assessment(FMA)_Health Status Chronic Stroke
Description: Upper extremity The total score means that severe <20, 20=<moderate<60, 60=<mild. Higher scores on the Fugl-Meyer Assessment indicate better upper limb motor control with reduced synergistic patterns, while lower scores indicate stronger synergistic patterns due to spasticity
  1) Reflex activity_max 4 score, 2) Volitional movement within synergies_ max 18, 3) Volitional movement mixing synergies_ max 6, 4) Volitional movement with little or no synergy_ max 6, 5) Normal reflex activity_max 2, 6) Wrist movement_ max 10, 7) Hand movement with grasp_ max 14, 8) coordination/speed_max 6.
  * Shoulder, Elbow and Forearm
    1. Reflex activity
    2. Volitional movement within synergies
    3. Volitional movement mixing synergies
    4. Volitional movement with little or no synergy
    5. Normal reflex activity
  * Wrist
  * Hand
  * Coordination/Speed
  * Total score is 66 points
Time Frame: Baseline
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Modified Ashworth Scale_Stiffness of Chronic Stroke
Description: Scoring for Triceps
  * MAS 0: No increase in tone
  * MAS 1: slight increase in tone giving a catch when slight increase in muscle t-tone, manifested by the limb was moved in flexion or extension.
  * MAS 1+: slight increase in muscle tone, manifested by a catch followed by minimal resistance throughout (ROM )
  * MAS 2: more marked increase in tone but more marked increased in muscle tone through most limb easily flexed
  * MAS 3: considerable increase in tone, passive movement difficult
  * MAS 4: limb rigid in flexion or extension The Modified Ashworth Scale (MAS) ranges from 0 to 4, where higher scores indicate more severe spasticity/increased muscle tone. A score of 0 represents normal muscle tone, while 4 represents the most severe level of spasticity.
Time Frame: Baseline
Population: The population analyzed enrolled all participants with inclusion criteria between chronic stroke and healthy
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Chronic Stroke | Healthy
Number analyzed (Participants) | 35 | 61
units on a scale | 1 [0 to 2] | 0 [0 to 0]

ADVERSE EVENTS:
Description: It involved observation at a specific point in time without any intervention. All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Chronic Stroke | Healthy
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
the absence of randomization increased the risk of confounding bias.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-07-19): https://cdn.clinicaltrials.gov/large-docs/58/NCT05683158/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-19): https://cdn.clinicaltrials.gov/large-docs/58/NCT05683158/SAP_001.pdf
  • Informed Consent Form (2022-07-19): https://cdn.clinicaltrials.gov/large-docs/58/NCT05683158/ICF_002.pdf